CLINICAL TRIAL: NCT05734313
Title: Telemedicine-Delivered Unified Protocol for Cognitive Behavioral Therapy for Anxiety and Depression in Young Adults With Type 1 Diabetes
Brief Title: Telemedicine-Delivered Unified Protocol for Cognitive Behavioral Therapy for Anxiety and Depression
Acronym: UP-CBT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other); DexCom, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-14517
Record Dates: First submitted 2023-02-02; First posted 2023-02-17 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Diabetes; Type 1 Diabetes
Keywords: Diabetes; Type 1 Diabetes; Depression; Anxiety; Diabetes Distress; Diabetes Management; Diabetes Self-Care
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Depression; Anxiety Disorders | interventions — Cognitive Behavioral Therapy; Continuous Glucose Monitoring

STUDY DESIGN:
Intervention Model Description: There will be two arms in this trial, (1) The Unified Protocol for Cognitive Behavioral Therapy (UP-CBT) Intervention Arm paired with use of continuous glucose monitor (CGM) and (2) CGM only. The active comparison condition of CGM only allows for the evaluation of whether directly targeting emotional disorders with UP-CBT adds value beyond the state-of-the-art approach to glycemic management in Type 1 Diabetes. To the extent that the relationship between emotional disorders and diabetes is bidirectional, a common assumption across research studies in this area, the comparison condition should benefit anxiety and depression outcomes through improved glycemic control and diabetes self-management.
Who Masked: Outcomes Assessor
Masking Description: Trained clinical interviewers blind to treatment assignment will administer structured clinical interviews to assess primary outcomes of anxiety and depression symptom severity at each assessment. Time in Range will be calculated from CGM data by an analyst who is blind to assignment. Hemoglobin A1c (HbA1c) will be collected via mailed kits at each assessment and analyzed by a lab blind to assignment. Anxiety and Depression severity data will be measured longitudinally throughout the trial, at baseline, immediately post-intervention, and at 9- and 12-months post-randomization by independent assessors blind to the assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Unified Protocol for Cognitive Behavioral Therapy (UP-CBT) with Continuous Glucose Monitoring (Experimental): Participants randomized to this arm will receive the Unified Protocol for Cognitive Behavioral Therapy (UP-CBT), enhanced by review of Continuous Glucose Monitoring (CGM) data. Participants will wear study-supplied CGM for the first 6 months of their participation in the trial.
  Interventions: Behavioral: Unified protocol for cognitive behavioral therapy (UP-CBT); Device: Continuous Glucose Monitoring (CGM)
- Continuous Glucose Monitoring (CGM) Only (Active Comparator): Participants randomized to receive Continuous Glucose Monitoring (CGM) will continue to receive their usual care and will also wear CGM throughout the first 6 months of their participation in the trial.
  Interventions: Device: Continuous Glucose Monitoring (CGM)

INTERVENTIONS:
Behavioral: Unified protocol for cognitive behavioral therapy (UP-CBT) — UP-CBT consists of approximately 16 individual sessions of CBT, conducted over the course of approximately 20 weeks. The UP-CBT consists of 5 core modules targeting negative emotionality and aversive reactions to emotional experiences. These modules are preceded by an introductory session that reviews the patient's presenting symptoms and provides a therapeutic rationale, as well as a module on motivational enhancement. The final module consists of relapse prevention. UP-CBT sessions will integrate a review of Continuous Glucose Monitoring (CGM) data and feedback will be provided by the therapist.
  Arms: Unified Protocol for Cognitive Behavioral Therapy (UP-CBT) with Continuous Glucose Monitoring
Device: Continuous Glucose Monitoring (CGM) — Use of commercially available, FDA-approved continuous glucose monitoring (CGM) for 6 months post-randomization. Usual diabetes care will continue and participants can initiate a CGM review from their healthcare providers, as desired. In addition, a nurse practitioner with expertise in CGM will train each participant via video recordings in the proper placement of the device, and technical issues, and provide basic teaching at the beginning of the trial on interpretation of CGM data and self-titration of insulin/self-management. Written materials and online resources for recognizing and managing anxiety and depressive disorders, along with self-management information and treatment options to discuss with providers will also be provided.

SUMMARY:
This project will evaluate a telemedicine-delivered, Unified Protocol for Cognitive-Behavioral Therapy (UP-CBT) enhanced with continuous glucose monitor (CGM) review to target anxiety and depressive symptoms and glycemic control in adults with type 1 diabetes.

DETAILED DESCRIPTION:
The efficacy of the Unified Protocol for Cognitive Behavioral Therapy (UP-CBT) combined with commercial FDA-approved Continuous Glucose Monitoring (CGM) will be tested in comparison to CGM only in a randomized controlled clinical trial. The central hypothesis is that the addition of the UP-CBT intervention will yield clinically significant improvements in anxiety and depressive symptom severity and glycemic control relative to CGM alone. We will recruit 94 adults (age 18-64) with suboptimally controlled type 1 diabetes and an anxiety or depressive disorder from a national population for an entirely virtual 12-month study over five years, with targeted recruitment of racial/ethnic minorities. In addition to standard measurement of hemoglobin A1c (HbA1c) for glycemic control and validated patient-reported outcome (PRO) surveys, the study integrates momentary psychological and behavioral data via smartphone-based ecological momentary assessment (EMA) with CGM data to assess day-to-day changes in affect, self-management, and glycemia over the course of the trial.

Qualitative information will be collected from people with Type 1 Diabetes (T1D) ages 35-64 to solicit suggestions and inform future study decisions. We will create 2-4 focus groups to ask their impressions about our current study and to explore key factors like establishing adult care and attending medical appointments, disease self-management, and adjusting to chronic disease. We will compare interview responses from participant groups who have high vs. low social needs and poor vs. good glycemic control.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes (T1D) duration ≥ 6 months
* 18-64 years old
* English- or Spanish-speaking
* Anxiety or depressive mood disorder as per structured diagnostic interview.

Exclusion Criteria:

* Developmental or sensory disability interfering with participation
* Current pregnancy
* Bipolar disorders, psychotic disorders, severe eating disorders, severe substance abuse disorders, or acute suicidal risk or self-harm
* Use of medications or recent medical procedures that would impact glycemic control or use of continuous glucose monitoring (CGM) over the study
* Received cognitive behavioral therapy (CBT) in last year or plans to initiate CBT; (6) temporary exclusion for recent initiation of psychotropic medication - must be on a stable dose for 6 weeks prior to enrollment.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 94 (Estimated)
Dates: Start 2023-03-31 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Anxiety symptom severity | Baseline and midway through treatment (3 months), immediately post-treatment (5.5 months) and 9- and 12- months post-baseline
  Participant ratings will be conducted via video conference by clinicians blinded to the condition, using the Structured Interview Guide for the Hamilton Anxiety Rating Scales (SIGH-A). SIGH-A measures the severity of a patient's somatic and psychic anxiety based on 14 parameters including anxious mood, tension, fears, insomnia, somatic complaints and behavior at the interview. Each item is assigned a 5-point score ranging from 0 (not present) to 4 (severe) yielding an overall possible score of 0-56. Higher SIGH-A scores denote increased severity of anxiety.
Depressive symptom severity | Baseline and midway through treatment (3 months), immediately post-treatment (5.5 months) and 9- and 12- months post-baseline
  Participant ratings will be conducted via video conference by clinicians blinded to the condition, using the Structured Interview Guide for the Hamilton Depression Rating Scales (SIGH-D). SIGH-D is a 29-item clinical interview that expands the 21-item Hamilton Depression Rating Scale for Depression (HAM-D) to include eight items assessing "atypical symptoms" of depression. Ranges for individual parameters vary but a score of 0 signifies less severity (e.g., no/absent) and incrementally higher scores represent more severe symptoms. Total SIGH-D scores can range from 0 to 90. A higher overall SIGH-D score denotes increased severity of Depression.

SECONDARY OUTCOMES:
Time in Range (TIR) calculated from Continuous Glucose Monitoring (CGM) | 6 months
  The percentage of time glucose values were within range (i.e., between 70-180 mg/dL) will be calculated from CGM data during the 6 months after randomization. Results will be summarized by study arm using basic descriptive statistics.
Hemoglobin A1c (HbA1c) | 6 months
  Hemoglobin A1c (HbA1c) values will be calculated using mailed point-of-care (POC) kits for home collection. Samples will be collected, returned, processed, and shipped for analysis by a central laboratory. HbA1c results will be summarized by study arm using basic descriptive statistics.

OTHER OUTCOMES:
Hemoglobin A1c (HbA1c) | 9 months
  Hemoglobin A1c (HbA1c) values will be calculated using mailed point-of-care (POC) kits for home collection. Samples will be collected, returned, processed, and shipped for analysis by a central laboratory. HbA1c results will be summarized by study arm using basic descriptive statistics.
Hemoglobin A1c (HbA1c) | 12 months
  Hemoglobin A1c (HbA1c) values will be calculated using mailed point-of-care (POC) kits for home collection. Samples will be collected, returned, processed, and shipped for analysis by a central laboratory. HbA1c results will be summarized by study arm using basic descriptive statistics.
Depressive symptom severity | 9 months
  Participant ratings will be conducted via video conference by clinicians blinded to the condition, using the Structured Interview Guide for the Hamilton Depression Rating Scales (SIGH-D). SIGH-D is a 29-item clinical interview that expands the 21-item Hamilton Depression Rating Scale for Depression (HAM-D) to include eight items assessing "atypical symptoms" of depression. Ranges for individual parameters vary but a score of 0 signifies less severity (e.g., no/absent) and incrementally higher scores represent more severe symptoms. Total SIGH-D scores can range from 0 to 90. A higher overall SIGH-D score denotes increased severity of Depression.
Depressive symptom severity | 12 months
  Participant ratings will be conducted via video conference by clinicians blinded to the condition, using the Structured Interview Guide for the Hamilton Depression Rating Scales (SIGH-D). SIGH-D is a 29-item clinical interview that expands the 21-item Hamilton Depression Rating Scale for Depression (HAM-D) to include eight items assessing "atypical symptoms" of depression. Ranges for individual parameters vary but a score of 0 signifies less severity (e.g., no/absent) and incrementally higher scores represent more severe symptoms. Total SIGH-D scores can range from 0 to 90. A higher overall SIGH-D score denotes increased severity of Depression.
Anxiety symptom severity | 9 months
  Participant ratings will be conducted via video conference by clinicians blinded to the condition, using the Structured Interview Guide for the Hamilton Anxiety Rating Scales (SIGH-A). SIGH-A measures the severity of a patient's somatic and psychic anxiety based on 14 parameters including anxious mood, tension, fears, insomnia, somatic complaints and behavior at the interview. Each item is assigned a 5-point score ranging from 0 (not present) to 4 (severe) yielding an overall possible score of 0-56. Higher SIGH-A scores denote increased severity of anxiety.
Anxiety symptom severity | 12 months
  Participant ratings will be conducted via video conference by clinicians blinded to the condition, using the Structured Interview Guide for the Hamilton Anxiety Rating Scales (SIGH-A). SIGH-A measures the severity of a patient's somatic and psychic anxiety based on 14 parameters including anxious mood, tension, fears, insomnia, somatic complaints and behavior at the interview. Each item is assigned a 5-point score ranging from 0 (not present) to 4 (severe) yielding an overall possible score of 0-56. Higher SIGH-A scores denote increased severity of anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Gonzalez, PhD, Principal Investigator — Albert Einstein College of Medicine
Locations (2):
- United States (2):
  - Boston University, Boston, Massachusetts
  - Albert Einstein College of Medicine, The Bronx, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Young-Hyman D, de Groot M, Hill-Briggs F, Gonzalez JS, Hood K, Peyrot M. Psychosocial Care for People With Diabetes: A Position Statement of the American Diabetes Association. Diabetes Care. 2016 Dec;39(12):2126-2140. doi: 10.2337/dc16-2053. No abstract available. PMID 27879358
- [Background] Gonzalez JS, Hood KK, Esbitt SA, Mukherji S, Kane NS, Jacobson A. Psychiatric and Psychosocial Issues Among Individuals Living With Diabetes. In: Cowie CC, Casagrande SS, Menke A, Cissell MA, Eberhardt MS, Meigs JB, Gregg EW, Knowler WC, Barrett-Connor E, Becker DJ, Brancati FL, Boyko EJ, Herman WH, Howard BV, Narayan KMV, Rewers M, Fradkin JE, editors. Diabetes in America. 3rd edition. Bethesda (MD): National Institute of Diabetes and Digestive and Kidney Diseases (US); 2018 Aug. CHAPTER 33. Available from http://www.ncbi.nlm.nih.gov/books/NBK567974/ PMID 33651537
- [Background] American Psychiatric Association. Diagnostic and statistical manual of mental disorders (5th ed.). 2013.
- [Background] Ellard KK, Fairholme CP, Boisseau CL, Farchione TJ, Barlow DH. Unified Protocol for the Transdiagnostic Treatment of Emotional Disorders: Protocol Development and Initial Outcome Data. Cogn Behav Pract. 2010 Feb;17(1):88-101. doi: 10.1016/j.cbpra.2009.06.002. Epub 2010 Jan 29. PMID 33762811
- [Background] Farchione TJ, Fairholme CP, Ellard KK, Boisseau CL, Thompson-Hollands J, Carl JR, Gallagher MW, Barlow DH. Unified protocol for transdiagnostic treatment of emotional disorders: a randomized controlled trial. Behav Ther. 2012 Sep;43(3):666-78. doi: 10.1016/j.beth.2012.01.001. Epub 2012 Jan 18. PMID 22697453
- [Background] Sakiris N, Berle D. A systematic review and meta-analysis of the Unified Protocol as a transdiagnostic emotion regulation based intervention. Clin Psychol Rev. 2019 Aug;72:101751. doi: 10.1016/j.cpr.2019.101751. Epub 2019 Jun 25. PMID 31271848
- [Background] Steele SJ, Farchione TJ, Cassiello-Robbins C, Ametaj A, Sbi S, Sauer-Zavala S, Barlow DH. Efficacy of the Unified Protocol for transdiagnostic treatment of comorbid psychopathology accompanying emotional disorders compared to treatments targeting single disorders. J Psychiatr Res. 2018 Sep;104:211-216. doi: 10.1016/j.jpsychires.2018.08.005. Epub 2018 Aug 3. PMID 30103069
- [Background] Cassiello-Robbins C, Southward MW, Tirpak JW, Sauer-Zavala S. A systematic review of Unified Protocol applications with adult populations: Facilitating widespread dissemination via adaptability. Clin Psychol Rev. 2020 Jun;78:101852. doi: 10.1016/j.cpr.2020.101852. Epub 2020 Apr 20. PMID 32360953
- [Background] Carlucci L, Saggino A, Balsamo M. On the efficacy of the unified protocol for transdiagnostic treatment of emotional disorders: A systematic review and meta-analysis. Clin Psychol Rev. 2021 Jul;87:101999. doi: 10.1016/j.cpr.2021.101999. Epub 2021 Mar 9. PMID 34098412
- [Background] Peters A, Laffel L; American Diabetes Association Transitions Working Group. Diabetes care for emerging adults: recommendations for transition from pediatric to adult diabetes care systems: a position statement of the American Diabetes Association, with representation by the American College of Osteopathic Family Physicians, the American Academy of Pediatrics, the American Association of Clinical Endocrinologists, the American Osteopathic Association, the Centers for Disease Control and Prevention, Children with Diabetes, The Endocrine Society, the International Society for Pediatric and Adolescent Diabetes, Juvenile Diabetes Research Foundation International, the National Diabetes Education Program, and the Pediatric Endocrine Society (formerly Lawson Wilkins Pediatric Endocrine Society). Diabetes Care. 2011 Nov;34(11):2477-85. doi: 10.2337/dc11-1723. No abstract available. PMID 22025785
- [Background] Srinivas P, Bodke K, Ofner S, Keith NR, Tu W, Clark DO. Context-Sensitive Ecological Momentary Assessment: Application of User-Centered Design for Improving User Satisfaction and Engagement During Self-Report. JMIR Mhealth Uhealth. 2019 Apr 3;7(4):e10894. doi: 10.2196/10894. PMID 30942698
- [Background] Yang YS, Ryu GW, Choi M. Methodological Strategies for Ecological Momentary Assessment to Evaluate Mood and Stress in Adult Patients Using Mobile Phones: Systematic Review. JMIR Mhealth Uhealth. 2019 Apr 1;7(4):e11215. doi: 10.2196/11215. PMID 30932866
- [Background] Miller KM, Foster NC, Beck RW, Bergenstal RM, DuBose SN, DiMeglio LA, Maahs DM, Tamborlane WV; T1D Exchange Clinic Network. Current state of type 1 diabetes treatment in the U.S.: updated data from the T1D Exchange clinic registry. Diabetes Care. 2015 Jun;38(6):971-8. doi: 10.2337/dc15-0078. PMID 25998289
- [Background] Livingstone SJ, Levin D, Looker HC, Lindsay RS, Wild SH, Joss N, Leese G, Leslie P, McCrimmon RJ, Metcalfe W, McKnight JA, Morris AD, Pearson DW, Petrie JR, Philip S, Sattar NA, Traynor JP, Colhoun HM; Scottish Diabetes Research Network epidemiology group; Scottish Renal Registry. Estimated life expectancy in a Scottish cohort with type 1 diabetes, 2008-2010. JAMA. 2015 Jan 6;313(1):37-44. doi: 10.1001/jama.2014.16425. PMID 25562264
- [Background] Rhodes ET, Prosser LA, Hoerger TJ, Lieu T, Ludwig DS, Laffel LM. Estimated morbidity and mortality in adolescents and young adults diagnosed with Type 2 diabetes mellitus. Diabet Med. 2012 Apr;29(4):453-63. doi: 10.1111/j.1464-5491.2011.03542.x. PMID 22150528
- [Background] Dabelea D, Stafford JM, Mayer-Davis EJ, D'Agostino R Jr, Dolan L, Imperatore G, Linder B, Lawrence JM, Marcovina SM, Mottl AK, Black MH, Pop-Busui R, Saydah S, Hamman RF, Pihoker C; SEARCH for Diabetes in Youth Research Group. Association of Type 1 Diabetes vs Type 2 Diabetes Diagnosed During Childhood and Adolescence With Complications During Teenage Years and Young Adulthood. JAMA. 2017 Feb 28;317(8):825-835. doi: 10.1001/jama.2017.0686. PMID 28245334
- [Background] Bryden KS, Peveler RC, Stein A, Neil A, Mayou RA, Dunger DB. Clinical and psychological course of diabetes from adolescence to young adulthood: a longitudinal cohort study. Diabetes Care. 2001 Sep;24(9):1536-40. doi: 10.2337/diacare.24.9.1536. PMID 11522695
- [Background] Rodwell L, Romaniuk H, Nilsen W, Carlin JB, Lee KJ, Patton GC. Adolescent mental health and behavioural predictors of being NEET: a prospective study of young adults not in employment, education, or training. Psychol Med. 2018 Apr;48(5):861-871. doi: 10.1017/S0033291717002434. Epub 2017 Sep 6. PMID 28874224
- [Background] 2014 Diabetes Health Care Cost Institute Utilization Report. Health Care Cost Institute. Published 2014. Accessed October 3, 2021. https://healthcostinstitute.org/images/easyblog_articles/276/HCCI-2017-Health-Care-Cost-and-Utilization-Report-02.12.19.pdf
- [Background] Sequeira PA, Pyatak EA, Weigensberg MJ, Vigen CP, Wood JR, Ruelas V, Montoya L, Cohen M, Speer H, Clark S, Peters AL. Let's Empower and Prepare (LEAP): Evaluation of a Structured Transition Program for Young Adults With Type 1 Diabetes. Diabetes Care. 2015 Aug;38(8):1412-9. doi: 10.2337/dc14-2577. Epub 2015 Apr 23. PMID 25906787
- [Background] Pyatak EA, Carandang K, Vigen CLP, Blanchard J, Diaz J, Concha-Chavez A, Sequeira PA, Wood JR, Whittemore R, Spruijt-Metz D, Peters AL. Occupational Therapy Intervention Improves Glycemic Control and Quality of Life Among Young Adults With Diabetes: the Resilient, Empowered, Active Living with Diabetes (REAL Diabetes) Randomized Controlled Trial. Diabetes Care. 2018 Apr;41(4):696-704. doi: 10.2337/dc17-1634. Epub 2018 Jan 19. PMID 29351961
- [Background] Bakhach M, Reid MW, Pyatak EA, Berget C, Cain C, Thomas JF, Klingensmith GJ, Raymond JK. Home Telemedicine (CoYoT1 Clinic): A Novel Approach to Improve Psychosocial Outcomes in Young Adults With Diabetes. Diabetes Educ. 2019 Aug;45(4):420-430. doi: 10.1177/0145721719858080. Epub 2019 Jun 27. PMID 31244396
- [Background] Kessler RC, Ruscio AM, Shear K, Wittchen HU. Epidemiology of anxiety disorders. Curr Top Behav Neurosci. 2010;2:21-35. PMID 21309104
- [Background] Zimmerman M, Clark HL, Multach MD, Walsh E, Rosenstein LK, Gazarian D. Have Treatment Studies of Depression Become Even Less Generalizable? A Review of the Inclusion and Exclusion Criteria Used in Placebo-Controlled Antidepressant Efficacy Trials Published During the Past 20 Years. Mayo Clin Proc. 2015 Sep;90(9):1180-6. doi: 10.1016/j.mayocp.2015.06.016. Epub 2015 Aug 12. PMID 26276679
- [Background] Lorenzo-Luaces L, Zimmerman M, Cuijpers P. Are studies of psychotherapies for depression more or less generalizable than studies of antidepressants? J Affect Disord. 2018 Jul;234:8-13. doi: 10.1016/j.jad.2018.02.066. Epub 2018 Feb 27. PMID 29522947
- [Background] Simoni JM, Wiebe JS, Sauceda JA, Huh D, Sanchez G, Longoria V, Andres Bedoya C, Safren SA. A preliminary RCT of CBT-AD for adherence and depression among HIV-positive Latinos on the U.S.-Mexico border: the Nuevo Dia study. AIDS Behav. 2013 Oct;17(8):2816-29. doi: 10.1007/s10461-013-0538-5. PMID 23812892
- [Background] Allen LB, White KS, Barlow DH, Shear MK, Gorman JM, Woods SW. Cognitive-Behavior Therapy (CBT) for Panic Disorder: Relationship of Anxiety and Depression Comorbidity with Treatment Outcome. J Psychopathol Behav Assess. 2010 Jun;32(2):185-192. doi: 10.1007/s10862-009-9151-3. Epub 2009 Jul 24. PMID 20421906
- [Background] Tsao JC, Lewin MR, Craske MG. The effects of cognitive-behavior therapy for panic disorder on comorbid conditions. J Anxiety Disord. 1998 Jul-Aug;12(4):357-71. doi: 10.1016/s0887-6185(98)00020-6. PMID 9699119
- [Background] Barlow DH, Farchione TJ, Bullis JR, Gallagher MW, Murray-Latin H, Sauer-Zavala S, Bentley KH, Thompson-Hollands J, Conklin LR, Boswell JF, Ametaj A, Carl JR, Boettcher HT, Cassiello-Robbins C. The Unified Protocol for Transdiagnostic Treatment of Emotional Disorders Compared With Diagnosis-Specific Protocols for Anxiety Disorders: A Randomized Clinical Trial. JAMA Psychiatry. 2017 Sep 1;74(9):875-884. doi: 10.1001/jamapsychiatry.2017.2164. PMID 28768327
- [Background] Gonzalez JS, McCarl LA, Wexler D DD, Cagliero E, Delahanty L, Soper TD, Goldman V, Knauz R, Safren SA. Cognitive Behavioral Therapy for Adherence and Depression (CBT-AD) in Type 2 Diabetes. J Cogn Psychother. 2010 Nov 1;24(4):329-343. doi: 10.1891/0889-8391.24.4.329. PMID 23667294
- [Background] Safren SA, Gonzalez JS, Wexler DJ, Psaros C, Delahanty LM, Blashill AJ, Margolina AI, Cagliero E. A randomized controlled trial of cognitive behavioral therapy for adherence and depression (CBT-AD) in patients with uncontrolled type 2 diabetes. Diabetes Care. 2014;37(3):625-33. doi: 10.2337/dc13-0816. Epub 2013 Oct 29. PMID 24170758
- [Background] Targum SD, Sauder C, Evans M, Saber JN, Harvey PD. Ecological momentary assessment as a measurement tool in depression trials. J Psychiatr Res. 2021 Apr;136:256-264. doi: 10.1016/j.jpsychires.2021.02.012. Epub 2021 Feb 14. PMID 33621911
- [Background] Mulvaney SA, Vaala SE, Carroll RB, Williams LK, Lybarger CK, Schmidt DC, Dietrich MS, Laffel LM, Hood KK. A mobile app identifies momentary psychosocial and contextual factors related to mealtime self-management in adolescents with type 1 diabetes. J Am Med Inform Assoc. 2019 Dec 1;26(12):1627-1631. doi: 10.1093/jamia/ocz147. PMID 31529065
- [Background] Hermanns N, Scheff C, Kulzer B, Weyers P, Pauli P, Kubiak T, Haak T. Association of glucose levels and glucose variability with mood in type 1 diabetic patients. Diabetologia. 2007 May;50(5):930-3. doi: 10.1007/s00125-007-0643-y. Epub 2007 Mar 17. PMID 17370057
- [Background] Wagner J, Armeli S, Tennen H, Bermudez-Millan A, Wolpert H, Perez-Escamilla R. A daily study of stressors, continuously measured glucose, and diabetes symptoms in latinos with type 2 diabetes. J Behav Med. 2021 Feb;44(1):94-103. doi: 10.1007/s10865-020-00162-1. Epub 2020 Jun 3. PMID 32494976
- [Background] Skaff MM, Mullan JT, Almeida DM, Hoffman L, Masharani U, Mohr D, Fisher L. Daily negative mood affects fasting glucose in type 2 diabetes. Health Psychol. 2009 May;28(3):265-72. doi: 10.1037/a0014429. PMID 19450031
- [Background] Polonsky WH, Fortmann AL. The influence of time in range on daily mood in adults with type 1 diabetes. J Diabetes Complications. 2020 Dec;34(12):107746. doi: 10.1016/j.jdiacomp.2020.107746. Epub 2020 Oct 7. PMID 33077350
- [Background] Bullis JR, Fortune MR, Farchione TJ, Barlow DH. A preliminary investigation of the long-term outcome of the Unified Protocol for Transdiagnostic Treatment of Emotional Disorders. Compr Psychiatry. 2014 Nov;55(8):1920-7. doi: 10.1016/j.comppsych.2014.07.016. Epub 2014 Jul 22. PMID 25113056
- [Background] Markowitz SM, Carper MM, Gonzalez JS, Delahanty LM, Safren SA. Cognitive-behavioral therapy for the treatment of depression and adherence in patients with type 1 diabetes: pilot data and feasibility. Prim Care Companion CNS Disord. 2012;14(2):PCC.11m01220. doi: 10.4088/PCC.11m01220. Epub 2012 Mar 15. PMID 22943030
- [Background] Esbitt SA, Batchelder AW, Tanenbaum ML, Shreck E, Gonzalez JS. "Knowing That You're Not the Only One": Perspectives on Group-Based Cognitive-Behavioral Therapy for Adherence and Depression (CBT-AD) in Adults With Type 1 Diabetes. Cogn Behav Pract. 2015 Aug 1;22(3):393-406. doi: 10.1016/j.cbpra.2014.02.006. PMID 26279614
- [Background] Agarwal S, Kanapka LG, Raymond JK, Walker A, Gerard-Gonzalez A, Kruger D, Redondo MJ, Rickels MR, Shah VN, Butler A, Gonzalez J, Verdejo AS, Gal RL, Willi S, Long JA. Racial-Ethnic Inequity in Young Adults With Type 1 Diabetes. J Clin Endocrinol Metab. 2020 Aug 1;105(8):e2960-9. doi: 10.1210/clinem/dgaa236. PMID 32382736
- [Background] Agarwal S, Schechter C, Gonzalez J, Long JA. Racial-Ethnic Disparities in Diabetes Technology use Among Young Adults with Type 1 Diabetes. Diabetes Technol Ther. 2021 Apr;23(4):306-313. doi: 10.1089/dia.2020.0338. Epub 2020 Dec 1. PMID 33155826
- [Background] Agarwal S, Raymond JK, Schutta MH, Cardillo S, Miller VA, Long JA. An Adult Health Care-Based Pediatric to Adult Transition Program for Emerging Adults With Type 1 Diabetes. Diabetes Educ. 2017 Feb;43(1):87-96. doi: 10.1177/0145721716677098. Epub 2016 Nov 15. PMID 28118128
- [Background] Agarwal S, Hilliard M, Butler A. Disparities in Care Delivery and Outcomes in Young Adults With Diabetes. Curr Diab Rep. 2018 Jul 14;18(9):65. doi: 10.1007/s11892-018-1037-x. PMID 30008025
- [Background] Agarwal S, Cappola AR. Continuous Glucose Monitoring in Adolescent, Young Adult, and Older Patients With Type 1 Diabetes. JAMA. 2020 Jun 16;323(23):2384-2385. doi: 10.1001/jama.2020.7058. No abstract available. PMID 32543670
- [Background] Garvey KC, Foster NC, Agarwal S, DiMeglio LA, Anderson BJ, Corathers SD, Desimone ME, Libman IM, Lyons SK, Peters AL, Raymond JK, Laffel LM. Health Care Transition Preparation and Experiences in a U.S. National Sample of Young Adults With Type 1 Diabetes. Diabetes Care. 2017 Mar;40(3):317-324. doi: 10.2337/dc16-1729. Epub 2016 Dec 22. PMID 28007779
- [Background] Kahkoska AR, Shay CM, Crandell J, Dabelea D, Imperatore G, Lawrence JM, Liese AD, Pihoker C, Reboussin BA, Agarwal S, Tooze JA, Wagenknecht LE, Zhong VW, Mayer-Davis EJ. Association of Race and Ethnicity With Glycemic Control and Hemoglobin A1c Levels in Youth With Type 1 Diabetes. JAMA Netw Open. 2018 Sep 7;1(5):e181851. doi: 10.1001/jamanetworkopen.2018.1851. PMID 30370425
- [Background] Agarwal S, Jawad AF, Miller VA. A multivariate model exploring the predictive value of demographic, adolescent, and family factors on glycemic control in adolescents with type 1 diabetes. Pediatr Diabetes. 2016 Nov;17(7):500-508. doi: 10.1111/pedi.12331. Epub 2015 Oct 21. PMID 26486450
- [Background] Ehrenreich-May J, Rosenfield D, Queen AH, Kennedy SM, Remmes CS, Barlow DH. An initial waitlist-controlled trial of the unified protocol for the treatment of emotional disorders in adolescents. J Anxiety Disord. 2017 Mar;46:46-55. doi: 10.1016/j.janxdis.2016.10.006. Epub 2016 Oct 17. PMID 27771133
- [Background] Sauer-Zavala S, Boswell JF, Gallagher MW, Bentley KH, Ametaj A, Barlow DH. The role of negative affectivity and negative reactivity to emotions in predicting outcomes in the unified protocol for the transdiagnostic treatment of emotional disorders. Behav Res Ther. 2012 Sep;50(9):551-7. doi: 10.1016/j.brat.2012.05.005. Epub 2012 Jun 9. PMID 22738907
- [Background] Boswell JF, Farchione TJ, Sauer-Zavala S, Murray HW, Fortune MR, Barlow DH. Anxiety sensitivity and interoceptive exposure: a transdiagnostic construct and change strategy. Behav Ther. 2013 Sep;44(3):417-31. doi: 10.1016/j.beth.2013.03.006. Epub 2013 Apr 2. PMID 23768669
- [Background] Mohr DC, Ho J, Duffecy J, Reifler D, Sokol L, Burns MN, Jin L, Siddique J. Effect of telephone-administered vs face-to-face cognitive behavioral therapy on adherence to therapy and depression outcomes among primary care patients: a randomized trial. JAMA. 2012 Jun 6;307(21):2278-85. doi: 10.1001/jama.2012.5588. PMID 22706833
- [Background] Raymond JK, Berget CL, Driscoll KA, Ketchum K, Cain C, Fred Thomas JF. CoYoT1 Clinic: Innovative Telemedicine Care Model for Young Adults with Type 1 Diabetes. Diabetes Technol Ther. 2016 Jun;18(6):385-90. doi: 10.1089/dia.2015.0425. Epub 2016 May 19. PMID 27196443
- [Background] Sheehan DV, Lecrubier Y, Sheehan KH, Amorim P, Janavs J, Weiller E, Hergueta T, Baker R, Dunbar GC. The Mini-International Neuropsychiatric Interview (M.I.N.I.): the development and validation of a structured diagnostic psychiatric interview for DSM-IV and ICD-10. J Clin Psychiatry. 1998;59 Suppl 20:22-33;quiz 34-57. PMID 9881538
- [Background] Shear MK, Vander Bilt J, Rucci P, Endicott J, Lydiard B, Otto MW, Pollack MH, Chandler L, Williams J, Ali A, Frank DM. Reliability and validity of a structured interview guide for the Hamilton Anxiety Rating Scale (SIGH-A). Depress Anxiety. 2001;13(4):166-78. PMID 11413563
- [Background] Williams J, Link M, Rosenthal N, Terman M. Structured Interview Guide for the Hamilton Depression Rating Scale-Seasonal Affective Disorder Version (SIGH-SAD). New York: New York State Psychiatric Institute.1988.
- [Background] Polonsky WH, Anderson BJ, Lohrer PA, Welch G, Jacobson AM, Aponte JE, Schwartz CE. Assessment of diabetes-related distress. Diabetes Care. 1995 Jun;18(6):754-60. doi: 10.2337/diacare.18.6.754. PMID 7555499
- [Background] Weinger K, Butler HA, Welch GW, La Greca AM. Measuring diabetes self-care: a psychometric analysis of the Self-Care Inventory-Revised with adults. Diabetes Care. 2005 Jun;28(6):1346-52. doi: 10.2337/diacare.28.6.1346. PMID 15920050
- [Background] Johnson SU, Ulvenes PG, Oktedalen T, Hoffart A. Psychometric Properties of the General Anxiety Disorder 7-Item (GAD-7) Scale in a Heterogeneous Psychiatric Sample. Front Psychol. 2019 Aug 6;10:1713. doi: 10.3389/fpsyg.2019.01713. eCollection 2019. PMID 31447721
- [Background] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Background] Perera MJ, Brintz CE, Birnbaum-Weitzman O, Penedo FJ, Gallo LC, Gonzalez P, Gouskova N, Isasi CR, Navas-Nacher EL, Perreira KM, Roesch SC, Schneiderman N, Llabre MM. Factor structure of the Perceived Stress Scale-10 (PSS) across English and Spanish language responders in the HCHS/SOL Sociocultural Ancillary Study. Psychol Assess. 2017 Mar;29(3):320-328. doi: 10.1037/pas0000336. Epub 2016 Jun 9. PMID 27280744
- [Background] Geddes J, Wright RJ, Zammitt NN, Deary IJ, Frier BM. An evaluation of methods of assessing impaired awareness of hypoglycemia in type 1 diabetes. Diabetes Care. 2007 Jul;30(7):1868-70. doi: 10.2337/dc06-2556. Epub 2007 Apr 6. No abstract available. PMID 17416785
- [Background] Gonder-Frederick LA, Schmidt KM, Vajda KA, Greear ML, Singh H, Shepard JA, Cox DJ. Psychometric properties of the hypoglycemia fear survey-ii for adults with type 1 diabetes. Diabetes Care. 2011 Apr;34(4):801-6. doi: 10.2337/dc10-1343. Epub 2011 Feb 23. PMID 21346182
- [Background] Manzar MD, BaHammam AS, Hameed UA, Spence DW, Pandi-Perumal SR, Moscovitch A, Streiner DL. Dimensionality of the Pittsburgh Sleep Quality Index: a systematic review. Health Qual Life Outcomes. 2018 May 9;16(1):89. doi: 10.1186/s12955-018-0915-x. PMID 29743066
- [Background] Laffel LM, Kanapka LG, Beck RW, Bergamo K, Clements MA, Criego A, DeSalvo DJ, Goland R, Hood K, Liljenquist D, Messer LH, Monzavi R, Mouse TJ, Prahalad P, Sherr J, Simmons JH, Wadwa RP, Weinstock RS, Willi SM, Miller KM; CGM Intervention in Teens and Young Adults with T1D (CITY) Study Group; CDE10. Effect of Continuous Glucose Monitoring on Glycemic Control in Adolescents and Young Adults With Type 1 Diabetes: A Randomized Clinical Trial. JAMA. 2020 Jun 16;323(23):2388-2396. doi: 10.1001/jama.2020.6940. PMID 32543683
- [Background] Snijders T BR. Multilevel Modeling: An Introduction to Basic and Advanced Multilevel Modeling. Sage Publications; 1999.
- [Background] Bauer DJ, Preacher KJ, Gil KM. Conceptualizing and testing random indirect effects and moderated mediation in multilevel models: new procedures and recommendations. Psychol Methods. 2006 Jun;11(2):142-63. doi: 10.1037/1082-989X.11.2.142. PMID 16784335
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Hilliard ME, Minard CG, Marrero DG, de Wit M, Thompson D, DuBose SN, Verdejo A, Monzavi R, Wadwa RP, Jaser SS, Anderson BJ. Assessing Health-Related Quality of Life in Children and Adolescents with Diabetes: Development and Psychometrics of the Type 1 Diabetes and Life (T1DAL) Measures. J Pediatr Psychol. 2020 Apr 1;45(3):328-339. doi: 10.1093/jpepsy/jsz083. PMID 31665389